CLINICAL TRIAL: NCT06652958
Title: A Phase 1, Open-Label, Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VH4527079, Administered Either Intravenously or Subcutaneously to Healthy Adults and Persons With HIV
Brief Title: A Study to Assess the Safety and Pharmacokinetics of a Human Monoclonal Antibody (VH4527079) in Healthy Adults and Persons With HIV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 221877
Record Dates: First submitted 2024-09-27; First posted 2024-10-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); VH4527079; Monoclonal Antibody; Safety; Pharmacokinetics (PK); Healthy Adults; Persons with HIV (PWH)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Arm A, Cohort 1 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 1 (lowest dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 2 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 2 (low dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 3 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 3 (mid-low dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 4 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 4 (mid-high dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 5 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 5 (high dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 6 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 6 (max dose) by IV infusion.
  Interventions: Biological: VH4527079
- Arm A, Cohort 7 (Experimental): Healthy adult participants receive a single dose of VH4527079 Dose 1 (lowest dose) by SC injection.
  Interventions: Biological: VH4527079
- Arm B, Cohort 8 (Experimental): Healthy adult participants receive three doses of VH4527079 dose that is selected in Arm A, by IV infusion, separated by a time interval.
  Interventions: Biological: VH4527079
- Arm B, Cohort 9 (Experimental): Participants with HIV receive three doses of VH4527079 dose that is selected in Arm A, by IV infusion, separated by a time interval.
  Interventions: Biological: VH4527079

INTERVENTIONS:
Biological: VH4527079 — VH4527079 solution for injection or infusion will be administered either by SC injection or IV infusion respectively.

SUMMARY:
This study evaluates the safety, tolerability, and pharmacokinetics (PK) of a single dose administration of VH4527079 by subcutaneous (SC) injection or by intravenous (IV) infusion in healthy adult participants and multiple dose administration by IV infusion in healthy adult participants and in Persons with HIV (PWH).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive at the time of signing the informed consent.
* Participants who are overtly healthy based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants who are able to understand and comply with protocol requirements and timetables, instructions, and protocol-stated restrictions.
* • For Cohort 9 (PWH in Arm B), well controlled HIV on first-line INSTI-based oral antiretroviral therapy (ART) without history of virologic failure. HIV infection is documented by any licensed rapid HIV rest or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry.
* Body weight more than or equal to (>=)50.0 kg for men and >=45.0 kg for women and Body Mass Index (BMI) within the range 18.5 to 31.0 kg/m^2.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  - Participants who are female at birth are eligible to participate if at least one of the following conditions applies: Not pregnant or breastfeeding and, at least, one of the following conditions apply:
  * Is not a Participant of childbearing potential (POCBP). OR
  * Is a POCBP and agrees to use a highly effective contraceptive method 3 weeks prior to the start of this study and during the study.
* Capable of giving signed informed consent.
* Willing to have samples stored for future research for participants in Arm B; Cohort 8 (Healthy Volunteers) and Cohort 9 (PWH in Arm B).

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders, or any medical condition capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Weight >115.0 kg.
* Any medical condition that is not well controlled.
* Positive HIV testing for participants enrolled in Arm A, Arm B Cohort 8, and Arm C.
* Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence during the study.
* The participant has an underlying skin disease or disorder, piercing, or tattoos that would interfere with assessment of injection site reactions (ISRs).
* History of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions.
* Any condition which, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to take oral medication.
* Unstable liver disease, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease).
* Known history of cirrhosis with or without viral hepatitis co-infection.
* History of clinically relevant hepatitis within last 6 months.
* For Cohort 9 (PWH in Arm B), untreated syphilis infection (i.e., positive syphilis testing at screening) without documentation of treatment. Participants who have successfully completed treatment at least 7 days previously are eligible if recruitment is open. Positive syphilis testing at screening for any other Cohort is exclusionary.
* Lymphoma, leukemia, or any malignancy (except for breast cancer) within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Participants who poses a significant suicidality risk.
* Any pre-existing physical or mental condition which, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome or sudden cardiac death. Any significant arrhythmia or ECG finding which, will interfere with the safety for the individual participant.
* Exposure to an experimental drug, human blood product, anticoagulants, or experimental vaccine (which does not have emergency, conditional, or standard market authorization) within 30 days, or within 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study intervention or plans to receive live vaccines during the study.
* Any previous use of HIV Pre-exposure prophylaxis (PrEP) or Post-exposure prophylaxis (PEP) in Arm A (Cohorts 1 through 7) or Arm B (Cohort 8 only), or Arm C (Cohorts 10-14) either oral or parenteral, is exclusionary.
* Any previous use of Neonatal Fc receptor blockers (e.g., efgartigimod alfa-fcab).
* The participant has ever received an investigational HIV vaccine.
* Any approved or experimental non-HIV vaccination (e.g., SARS-CoV-2, HBV, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment (Day 0).
* Exposure to an experimental drug, human blood product, anticoagulants or vaccine (which does not have emergency, conditional, or standard market authorization) within 30 days, or within 5 half-lives of the test agents, or twice the duration of the biological effect of the test agents, whichever is longer, prior to the first dose of study treatment or plans to receive live vaccines during the study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities or vaccines within 12 months prior to the first dosing day.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing.
* Participants who require concomitant medications known to be associated with a prolonged QTc.
* Participants receiving any protocol-prohibited medication(s) and who are unwilling or unable to switch to an alternate medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) of Grade 2 and above severity | Up to Week 24 follow-up period
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of AEs will be assessed using Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life threatening and Grade 5=Death.
Area under the plasma-concentration time curve from time zero to infinity (AUC0-inf) of VH4527079 | From Day 1 Up to Week 24 follow-up period
Area under the plasma-concentration time curve from time zero to the last quantifiable concentration (AUC0-tlast) of VH4527079 | From Day 1 Up to Week 24 follow-up period
Area under the plasma-concentration time curve from defined interval between doses (AUCtau) of VH4527079 | From Day 1 Up to Week 24 follow-up period
Maximum observed plasma concentration (Cmax) of VH4527079 | From Day 1 Up to Week 24 follow-up period
Time to maximum observed plasma concentration (Tmax) of VH4527079 | From Day 1 Up to Week 24 follow-up period
Apparent terminal half-life (t1/2) of VH4527079 | From Day 1 Up to Week 24 follow-up period

SECONDARY OUTCOMES:
AUC0-inf of VH4527079 after a single dose administered via SC route relative to IV administration | From Day 1 Up to Week 24 follow-up period
AUC0-tlast of VH4527079 after a single dose administered via SC route relative to IV administration | From Day 1 Up to Week 24 follow-up period
Cmax of VH4527079 after a single dose administered via SC route relative to IV administration | From Day 1 Up to Week 24 follow-up period
Post-baseline values for chemistry panels: Glucose (fasting), Blood Urea Nitrogen, Creatinine, Calcium, Magnesium, Potassium, Phosphate, Direct Bilirubin, Total Bilirubin and Fasting lipid panel (milligrams per deciliter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
  Fasting lipid panel included cholesterol, triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL)
Post-baseline values for chemistry panels: AST/SGOT, ALT/SGPT, ALP and CPK (International Units per liter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
  Chemistry panels included Aspartate aminotransferase (AST)/ Serum glutamic-oxalo-acetic transaminase (SGOT), Alanine aminotransferase (ALT)/ Serum glutamic-pyruvic transaminase (SGPT), Alkaline phosphatase (ALP) and Creatinine phosphokinase (CPK)
Post-baseline values for chemistry panels: Amylase and Lipase (fasting) (Units per Liter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for chemistry panels: Total Protein (Grams per deciliter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for chemistry panels: Sodium chloride and Bicarbonate (milliequivalents per liter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Platelet count (cells per microliter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Red Blood Cell (RBC) Count (million cells per microliter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Hemoglobin (Hgb) (grams per deciliter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Hematocrit (Proportion of red blood cells in blood) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Mean Corpuscular Volume (MCV) (Femtoliters) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Mean Corpuscular Hemoglobin (MCH) (Picograms) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Reticulocytes (Percentage of reticulocytes) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for hematology panels: Differential count of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per liter) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for coagulation panels: Prothrombin time (PT) and Partial Thromboplastin Time (PTT) (Seconds) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Post-baseline values for coagulation panels: International normalized ratio (INR) (Ratio) | From Day 1 (pre-Dose 1) Up to Week 24 follow-up period
Change from baseline values for chemistry panels: Glucose (fasting), Blood Urea Nitrogen, Creatinine, Calcium, Magnesium, Potassium, Phosphate, Direct Bilirubin, Total Bilirubin and Fasting lipid panel (milligrams per deciliter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
  Fasting lipid panel included cholesterol, triglycerides, HDL, LDL
Change from baseline values for chemistry panels: AST/ SGOT, ALT/ SGPT, ALP and CPK (International Units per liter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for chemistry panels: Amylase and Lipase (fasting) (Units per Liter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for chemistry panels: Total Protein (Grams per deciliter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for chemistry panels: Sodium chloride and Bicarbonate (milliequivalents per liter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: Platelet count (cells per microliter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: RBC Count (million cells per microliter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: Hgb (grams per deciliter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: Hematocrit (Proportion of red blood cells in blood) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: MCV (Femtoliters) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: MCH (Picograms) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: Reticulocytes (Percentage of reticulocytes) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for hematology panels: Differential count of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per liter) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for coagulation panels: PT and PTT (Seconds) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Change from baseline values for coagulation panels: INR (Ratio) | From Day 1 (pre-Dose 1) up to Week 24 follow-up period
Number of participants with maximum post-baseline QT interval corrected (QTc) values compared to baseline by category | Up to Week 24 follow-up period
  QTc values will be categorized as no change= number of participants with QTc values less than or equal to (<=)450 milliseconds (msec), any increase= number of participants with QTc values more than (>)450 - 480 msec, number of participants with QTc values >480 -500 msec, and number of participants with QTc values >500 msec
Number of participants with maximum post-baseline increases in QTc values compared to baseline by category | Up to Week 24 follow-up period
  Post-baseline increase in QTc values will be categorized by number of participants with QTc value increase of <=30 msec, number of participants with QTc value increase of 31 - 60 msec, and number of participants with QTc value increase of >60 msec
Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline for diastolic and systolic blood pressure | Up to Week 24 follow-up period
  Number of participants with post-baseline changes will be categorized as change to low, change to within range or no change, and change to high
Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline for pulse rate | Up to Week 24 follow-up period
  Number of participants with post-baseline changes will be categorized as change to low, change to within range or no change, and change to high
Number of participants with any AEs and AEs by severity | Up to Week 24 follow-up period
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of AEs will be assessed using Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life threatening and Grade 5=Death.
Number of participants who discontinue treatment due to AEs | Up to Week 24 follow-up period

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf